CLINICAL TRIAL: NCT06241885
Title: The Effect of Gynaecological Drape and Specially Developed Gynaecological Shorts on Anxiety, Pain, and Satisfaction Related to First Vaginal Examination in Women: a Randomised Controlled Study
Brief Title: Anxiety, Pain, and Satisfaction Related to First Vaginal Examination in Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Deniz Akyıldız, Assoc. Prof. Dr., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: First Vaginal Examination
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Anxiety; Pain; Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Pain; Personal Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group I (Experimental): Women in Intervention Group II will wear gynaecological shorts specially developed by the researchers before vaginal examination. These shorts will be made of disposable fabric and will be sewn by the researchers in four different sizes (S-M-L-XL) according to the weight of the women. The middle part of the shorts to be developed will be closed with a snap button, and the opening will be provided when the snap button is opened during vaginal examination. In addition, these shorts will be approximately knee-cap length for women.
  Interventions: Behavioral: Intervention group I
- Control (No Intervention): The women in the control group will not be subjected to any additional hospital procedure during vaginal examination. Privacy curtains are routinely used in the hospital.

INTERVENTIONS:
Behavioral: Intervention group I — Women in Intervention Group II will wear gynaecological shorts specially developed by the researchers before vaginal examination. These shorts will be made of disposable fabric and will be sewn by the researchers in four different sizes (S-M-L-XL) according to the weight of the women. The middle part of the shorts will be closed with a snap button, and the opening will be provided when the snap button is opened during vaginal examination. In addition, these shorts will be approximately knee-cap length for women.
  Arms: Intervention group I

SUMMARY:
The Effect of Gynaecological Drape and Specially Developed Gynaecological Shorts on Anxiety, Pain and Satisfaction Related to First Vaginal Examination in Women: A Randomised Controlled Study

DETAILED DESCRIPTION:
Many women feel anxiety and pain about gynecological examination. The aim of the study was to investigate the effect of gynaecological drape and specially developed gynaecological shorts used for the first time in vaginal examination on anxiety, pain and satisfaction related to examination.

ELIGIBILITY:
Inclusion Criteria:

* Literate,
* 18 years of age or older,
* Can speak and understand Turkish,
* You are a woman who is having a vaginal examination for the first time
* Women who volunteered to participate in the study

Exclusion Criteria:

* Physical or mental illness that prevents them from communicating,
* Vaginal examination by a health professional other than the designated gynaecologist,
* Those who answered the research questions incompletely and
* Women who want to withdraw from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 10 minutes before and 10 minutes after vaginal examination
  Anxiety levels of women related to vaginal examination will be measured using The Trait Anxiety Inventory Form in intervention I, II, and control group.
Pain level | 10 minutes before and 10 minutes after vaginal examination
  Pain levels of women related to vaginal examination will be measured using VAS Pain Scale in intervention I, II, and control group.
Satisfaction level | 10 minutes after vaginal examination
  It will be used to assess women's satisfaction with vaginal examination. In this scale, women will be asked to indicate the level of satisfaction from 1 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No